CLINICAL TRIAL: NCT02074826
Title: Analysis of the Interplay Between Genetic Risk Variants for Atrial Fibrillation and Pathological Changes That Associate With the Disease
Brief Title: Left Atrial Low vOltage Zone, GenetIC Markers and Outcomes in Patients After Atrial Fibrillation abLation
Acronym: LOGICAL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Technische Universität Dresden (Other)
Collaborators: Landspitali University Hospital (Other)
Responsible Party: Principal Investigator, Mathias Forkmann, Dr. med., Technische Universität Dresden
Other Study IDs: GEN-AFIB-REG
Record Dates: First submitted 2014-02-27; First posted 2014-02-28 (Estimated); Last update posted 2015-02-13 (Estimated); Status verified 2015-02

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Blood samples in EDTA plastic vaccutainers will be collected from the study participants for genetic testing
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Atrial fibrillation: * Genotyping of the AF associated variants
  * Measurement of the amount of left atrial fibrosis

SUMMARY:
This prospective, single-centre cohort study aims to investigate the association between known genetic Atrial Fibrillation (AF) risk variants and the amount of left atrial fibrosis found in patients undergoing clinically indicated AF catheter ablation procedures.

Left atrial fibrosis is increasingly recognized as a fundamental part of the pathomorphological substrate creating an electrophysiological environment needed for electrical conduction heterogeneities. Such identification and treatment of left atrial fibrosis has already entered routine clinical use for RF catheter ablation in an attempt to develop an individualized and tailored treatment strategy. Today, it is unclear what impacts the development, the extent and the localization of left atrial fibrosis in different patients.

A number of genetic risk variants have been described that confer risk of AF and have been widely replicated. This indicates that genetic variants contribute to the risk of the individual to develop AF throughout his life. However, the mechanisms of how genetic variant impact the development of clinical arrhythmias is not yet well understood.

We hypothesize that genetic influences that lead to tissue changes may play a role in the development of the arrhythmia substrate for AF. This is likely to be especially true for those with a relatively brief history of AF and modest clinical disease burden. Therefore, we plan to investigate the association between known genetic AF variants and a detailed disease phenotype obtained from individual left atrial voltage mapping.

DETAILED DESCRIPTION:
The patient is referred for a radiofrequency (RF) ablation procedure for AF on clinical indications. All patients undergoing this procedure and fulfilling the inclusion criteria and not having any exclusion criteria are invited to participate in the study. After written informed consent, a patient is subjected to the study protocol of AF ablation. Detailed clinical information is obtained in addition to all data from imaging studies.

For genetic testing blood samples in EDTA (ethylenediaminetetraacetic) vacutainers will be collected from the study participants that will be performed at deCODE genetics in Reykjavik, Iceland. Samples will be frozen at -20°C and shipped to deCODE (deCODE genetics, Sturlugata 8, IS-101 Reykjavik, Iceland) in batches on ice. All sample handling, DNA isolation, and genotyping at deCODE will be performed in Clinical Laboratory Improvement Amendments (CLIA) and College of American Pathologists (CAP) accredited laboratories. The blood samples collected will be labelled using stickers with encrypted identifiers provided by deCODE. The key linking encrypted identifiers and the patient names will be stored in a secure location by the primary investigator in Dresden, Germany. The clinical data sent to deCODE will be encrypted in the same manner. Neither participants or third parties (e.g. health care insurance companies) will have any access to the genetic information collected.

Genotyping of the AF associated variants: DNA will be isolated in deCODE's CLIA and CAP accredited diagnostics laboratory from blood samples using the Chemagen method (Perkin Elmer). The SNPs (single nucleotide polymorphism) outlined in Table 1 will be genotyped using the Centaurus (Epoch Biosciences) platform. The genotyping of these markers have been analytically validated at deCODE using a comprehensive validated LIMS (Laboratory Information Management System) system that tracks every step in the process from registration to the final test report. Genotyping results for study participants will be stored in deCODE database under encrypted identifiers.

Prior to the ablation procedure, transesophageal echocardiography will be performed to exclude thrombus formation within the LA (left atrium). Electrophysiological studies are going to be performed in the post-absorptive state under deep sedation using midazolam and propofol. All antiarrhythmic medications will be discontinued at least five half-lives before the study, except amiodarone. Conventional 12-lead surface ECG (filtered 0.05-100 Hz) and bipolar intracardiac electrogram recordings (filtered 30-500 Hz) are amplified and displayed on Bard Laboratory System, (Bard Electrophysiology, Billerica, MA). A quadripolar and a decapolar catheter are introduced via the left femoral vein into the right ventricular apex and coronary sinus (CS) with a proximal pole at the CS ostium respectively. If atrial fibrillation (AF) is present in the beginning, a electric cardioversion (up to 3 times) will be performed to obtain sinus rhythm (SR).

A single transseptal puncture under fluoroscopic guidance will provide access into the LA. Repeated doses of heparin will be used to maintain an activated clotting time of 250 to 350 seconds throughout the whole procedure.

Mapping and ablation procedures will be guided by a 3D electroanatomical mapping system (CARTO 3, Biosense Webster, Inc., Diamond Bar, CA, USA or Ensite-Velocity, Endocardial Solutions, Inc., St. Paul, Minnesota, USA) in all patients. To quantify the amount of left atrial fibrosis, a bipolar voltage map will be carried out simultaneously during the CT-based 3D reconstruction of left atrium. All points will be taken in sinus rhythm. Radiofrequency alternating current will be delivered in a unipolar mode between the irrigated-tip electrode of the ablation catheter (Surround Flow, Biosense Webster or IBI Therapy CoolFlex, St. Jude Medical) and an external back plate electrode. The standard ablation settings include a preselected power of 40 W, and a flow rate of 15 or 17 ml/min (15 ml/min for Surround Flow, and 17 ml/min for CoolFlex). A temperature probe in the esophagus at the level of the LA is used to tag the esophageal location and to provide intraesophageal temperature feedback during the procedure. For the ablation procedure a ablation protocol is completed.

The following procedure data is recorded:

* Procedure date
* Initial rhythm: sinus rhythm, atrial fibrillation, atrial tachycardia
* Procedure time
* Fluoroscopy time and dose
* Ablation duration
* Ablation energy
* Isolation of each pulmonary vein
* Adverse events / procedure-related events: tamponade, stroke, myocardial infarction, pulmonary embolism, pulmonary edema

The primary end point is reached when a detailed endocardial voltage mapping has been performed and correlated with the suggested genetic AF markers.

ELIGIBILITY:
Inclusion Criteria:

* Documented atrial fibrillation in 12-lead ECG
* Paroxysmal or persistent symptomatic atrial fibrillation
* Ineffectiveness of antiarrhythmic medication (at least 1 medication) or indication for primary AF ablation according to current guidelines
* Age 18-75 years

Exclusion Criteria:

* Reversible etiology of atrial fibrillation
* Pregnancy
* Women of childbearing potential without a negative pregnancy test within 48 hours prior to the ablation procedure
* Known intracardiac or other thrombi
* Contraindication to anticoagulation
* Previous left atrial ablation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from our primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2014-03; Primary Completion 2016-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Association between the suggested genetic AF risk variants and the amount of left atrial low voltage zones | baseline
  The primary endpoint of the study measures the association between the suggested genetic AF risk variants and the amount of left atrial fibrosis found on detailed endocardial voltage mapping.

SECONDARY OUTCOMES:
Fluoroscopy exposure | baseline
Procedural ablation duration | baseline
Freedom from recurrences of AF or MRT (magnetic resonance tomography) after substrate guided AF ablation during follow up | 6 and 12 months after inclusion
Association between the proposed genetic markers and the patients clinical characteristics | baseline
Association between the proposed genetic markers and short and long term ablation success | 6 and 12 months afte inclusion
Association between the proposed genetic markers and hard clinical outcome parameters | 6 and 12 months after inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Piorkowski, PD, Study Chair — Department of Electrophysiology, University of Dresden - Heart Center; David O. Arnar, Dr, Study Chair — Department of Cardiology, Landspitali University Hospital Heart; Thomas P Gaspar, Dr., Principal Investigator — Department of Electrophysiology, University of Dresden - Heart Center; Mathias Forkmann, Dr., Principal Investigator — Department of Electrophysiology, University of Dresden - Heart Center
Locations (1):
- Heart Center Dresden, Depart. of Electrophysiology, Dresden, Germany